CLINICAL TRIAL: NCT06061627
Title: A Randomized Controlled Trial of Left Bundle brAnch opTimized Cardiac Resynchronization Therapy Versus conventionaL Bi-vEntricular Pacing in Heart Failure Patients With Nonspecific Intraventricular Conduction Delay
Brief Title: A Randomized Controlled Trial of LOT-CRT Versus conventionaL BiVP in Heart Failure Patients With NICD
Acronym: BATTLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Sir Run Run Shaw Hospital (Other); Fu Wai Hospital, Beijing, China (Other); West China Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The First People's Hospital of Yunnan (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Guangdong Provincial People's Hospital (Other); Shanghai Tong Ren Hospital (Other); Fujian Provincial Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FirstNanjingMU005
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Intraventricular Block
Keywords: Left bundle branch area pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOT-CRT group (Experimental): In this arm, an right artrial (RA) lead, an implantable cardioverter defibrillator (ICD) lead and a LV pacing lead are placed are conventionally implanted.
  A left bundle branch pacing(LBBP) lead is attempted to be placed.
  Interventions: Procedure: LOT-CRT group
- BiVP group (Active Comparator): In this arm, an RA lead , an ICD lead and a LV pacing lead are placed.
  Interventions: Procedure: BiVP group

INTERVENTIONS:
Procedure: LOT-CRT group — In addition to the leads implanted in BiVP group, it is also necessary to implant the left bundle branch area pacing(LBBAP) leads
  LBBAP includes LBBP and LVSP.
  LBBP is defined if fulfilling criterion 1 and at least one in criteria 2:
  1. Paced morphology of RBBD in surface lead V1 (QR, Qr, rSr', rSR' or Qrs);
  2. One of the following should be met, while the pacing threshold ≤ 1.5V/0.5ms:
     1. Selective LBBP capture pattern appears, with an iso-electrical window between the pacing spike and QRS onset;
     2. When reducing the output voltage, the LVAT undergoes a sudden change of>10ms;
  If criterion 1 is fulfilled but none in criteria 2 is met, the procedure is considered to be left ventricular septal pacing (LVSP).
  Arms: LOT-CRT group
Procedure: BiVP group — Implantation of a LV pacing lead is attempted using the standard-of-care technique first.
  Arms: BiVP group

SUMMARY:
BATTLE study has been designed as a prospective, multi-center, randomized, controlled trial. This study will enroll 83 patients with chronic heart failure accompanied by intraventricular block (NICD) over an estimated recruitment period of 3 years. An LOT-CRT group will be compared with a group of conventional BiVP in the follow-up of at least 6 months. The study aimed to compare the curative effect of LOT-CRT in preserving LV systolic function with traditional BiVP in chronic heart failure patients with NICD.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy is a standardized treatment strategy for patients with chronic heart failure complicated by wide QRS waves. With the continuous development of physiological pacing technology, traditional cardiac resynchronization therapy, namely biventricular pacing technology, is constantly challenged. Left bundle branch area pacing (LBBAP), as the main method of physiological pacing technology, is currently increasingly widely used in clinical practice. In recent years, research has mainly focused on heart failure patients with wide QRS waves such as non ischemic cardiomyopathy and typical left bundle branch block (LBBB). The recently published LBBP-RESYNC study was a randomized controlled study comparing left bundle branch pacing (LBBP) and biventricular pacing. The results showed that LBBP can achieve better improvement in left ventricular function compared to traditional biventricular pacing.

Compared with patients with typical LBBB, traditional biventricular pacing synchronized treatment is less effective in chronic heart failure patients accompanied by intraventricular block (NICD), which is closely related to the electrophysiological mechanism of LBBB. The blocking site of typical LBBB is generally located within the His bundle to the proximal end of the left bundle branch, while the distal end of the left bundle branch is relatively healthy. Therefore, LBBP can completely correct this type of LBBB and significantly narrow the QRS wave; The electrophysiological mechanism of NICD is relatively complex, and there may be multiple blocking sites, and LBBP cannot be completely corrected. How to improve the treatment efficacy and clinical prognosis of chronic heart failure patients with NICD is an important scientific issue that urgently needs to be solved. It is unclear whether left bundle branch pacing technology can provide support for cardiac function in such patients.

Traditional biventricular pacing combines right ventricular and left epicardial pacing; LBBAP combined with left ventricular epicardial pacing, also known as LOT-CRT, is an innovative pacing method. This study aims to explore the application value of LBBAP in patients with chronic heart failure and NICD.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or non ischemic cardiomyopathy
2. Optimal medical therapy for at lest 3 months
3. NYHA class II-IV
4. LVEF≤35% as assessed by echocardiography
5. Sinus rhythm (may have paroxysmal atrial fibrillation)
6. QRS duration ≥ 150ms
7. Intraventricular block (NICD), QRS morphology is neither LBBB nor RBBB

Exclusion Criteria:

1. Valvular heart disease that requires or has undergone surgical intervention
2. After mechanical tricuspid valve replacement
3. Persistent or permanent atrial fibrillation or atrial flutter
4. Second or third degree atrioventricular block
5. Have a history of acute myocardial infarction within 3 months prior to enrollment
6. Patient's expected survival time is less than 12 months
7. Pregnant or planned to conceive
8. Ventricular septal hypertrophy (ventricular septal thickness exceeds 15mm at the end of diastole)
9. Patients with simple and persistent left superior vena cava
10. Patients with existing pacemaker implantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction(LVEF) | Baseline; 6-month follow-up
  Changes from baseline LVEF(unit: %) assessed by echocardiography at follow-up

SECONDARY OUTCOMES:
Paced QRS duration | Postoperative day 1; 1-month,3-month and 6-month follow-up
  Paced QRS duration is evaluated postoperative day 1 and 1 months, 3 months and 6 months after implantation.
A combined clinical endpoint of all-cause mortality and heart failure hospitalization, | 6-month follow-up
  Including date and number of all-cause mortalityand heart failure hospitalization,
Left ventricular end systolic volume(LVESV) | Baseline; 3-month, 6-month follow-up
  Changes from baseline LVESV(unit: mL) assessed by echocardiography at follow-up
Left ventricular end diastolic volume(LVEDV) | Baseline; 3-month, 6-month follow-up
  Changes from baseline LVEDV(unit: mL) assessed by echocardiography at follow-up
Left ventricular end systolic diameter(LVESD) | Baseline; 3-month, 6-month follow-up
  Changes from baseline LVESD(unit: mm) assessed by echocardiography at follow-up
Left ventricular end diastolic diameter(LVEDD) | Baseline; 3-month, 6-month follow-up
  Changes from baseline LVEDD(unit: mm) assessed by echocardiography at follow-up
Change in Quality Of Life Questionnaire score between baseline and follow-up | Baseline; 3-month, 6-month follow-up
  Reflect the effect of cardiac funtion on quality of life, and higher scores represent a worse outcome
Changes in New York Heart Association Heart Function Classification between baseline and follow-up | Baseline; 3-month, 6-month follow-up
  The higher the classification, the more severe the heart failure symptoms(four levels: I, II, III and IV)
Changes in 6-minute Walk Distance between baseline and follow-up | Baseline; 3-month, 6-month follow-up
  Distance that a participant walk within 6 minutes
Changes in concentration of NT-proBNP in blood between baseline and follow-up | Baseline; 3-month, 6-month follow-up
  Blood test is performed at each time frame to determine the concentration of NT-proBNP(unit: pg/mL)
Incidence of stroke events | 6-month follow-up
  Including date and number of stroke
A combined arrhythmia endpoint of new-onset atrial fibrillation and malignant ventricular arrhythmia | 6-month follow-up
  Including date and number of new-onset atrial fibrillation and malignant ventricular arrhythmia
Success rate of LBBAP implantation Success rate of LBBAP implantation Success rate of LBBAP implantation Success rate of LBBAP implantation Success rate of LBBAP implantation | Operative day
  Success rate of LBBAP in LOT-CRT group

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Zou, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Yangang Su, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang Y, Zhu H, Hou X, Wang Z, Zou F, Qian Z, Wei Y, Wang X, Zhang L, Li X, Liu Z, Xue S, Qin C, Zeng J, Li H, Wu H, Ma H, Ellenbogen KA, Gold MR, Fan X, Zou J; LBBP-RESYNC Investigators. Randomized Trial of Left Bundle Branch vs Biventricular Pacing for Cardiac Resynchronization Therapy. J Am Coll Cardiol. 2022 Sep 27;80(13):1205-1216. doi: 10.1016/j.jacc.2022.07.019. PMID 36137670
- [Result] Jastrzebski M, Moskal P, Huybrechts W, Curila K, Sreekumar P, Rademakers LM, Ponnusamy SS, Herweg B, Sharma PS, Bednarek A, Rajzer M, Vijayaraman P. Left bundle branch-optimized cardiac resynchronization therapy (LOT-CRT): Results from an international LBBAP collaborative study group. Heart Rhythm. 2022 Jan;19(1):13-21. doi: 10.1016/j.hrthm.2021.07.057. Epub 2021 Jul 30. PMID 34339851